CLINICAL TRIAL: NCT00671593
Title: Genetics of Environmental Asthma: Differential Gene Expression in the Lung and Peripheral Blood After Inhaled Allergen Challenge
Brief Title: Differential Gene Expression in Lung and Peripheral Blood After Inhaled Allergen Challenge
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: funding terminated
Sponsor: John Sundy (Other)
Responsible Party: Sponsor-Investigator, John Sundy, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00008369; 8874-07-8R1 (Other: Duke Legacy ID); 12496-CP-005 (Other: NIEHS)
Record Dates: First submitted 2008-05-02; First posted 2008-05-05 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Atopic Asthma; Healthy
Keywords: Allergy; Asthma; healthy; Normal
MeSH Terms: conditions — Hypersensitivity; Asthma | interventions — Antigens, Dermatophagoides; Phenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental inhaled dust mite (Experimental): All subjects receive the same experimental inhaled challenge interventions
  Interventions: Biological: House Dust Mite; Biological: Diluent

INTERVENTIONS:
Biological: House Dust Mite — Dermatophagoides pteronyssinus: nebulized inhaled dosing is every 10 minutes per protocol limits at the following Allergen Concentration , (5 breaths of duration 0.8 seconds using a dosimeter) 0.0 AU, 0.3 AU/ml,
  1 AU/ml, 3 AU/ml, 10 AU/ml, 30 AU/ml, 100 AU/ml, 300 AU/ml, 1000 AU/ml, 3000 AU/ml
  Other Names: Allergen Extract Stand. Mite Dermatophagoides pteronyssinus
Biological: Diluent — Greer lab allergen extract diluent (0.5% sodium chloride, 0.25% sodium bicarbonate, 50% glycerin (v/v), and 0.4% phenol)nebulized inhaled dosing is every 10 minutes per protocol limits at the following Diluent Concentration, (5 breaths of duration 0.8 seconds using a dosimeter)
  Other Names: diluent(0.5% Nacl,0.25% NaHCO3,50% glycerin,& 0.4% phenol)

SUMMARY:
The purpose of this study is to identify the genes in important airway cells that are specifically expressed following inhalation of house dust mite allergen among study subjects with either allergic asthma or healthy normal phenotypes. This approach is designed to identify novel genes associated with both asthma pathogenesis (differentially expressed in the exposure-response study) and asthma susceptibility (genetically associated with asthma in a linkage/association study) for drug targets.

DETAILED DESCRIPTION:
The purpose of this study is to identify the genes in airway epithelial and BAL cells that are differentially expressed following inhalation of house dust mite allergen among study subjects with allergic asthma and normal phenotypes. This approach is designed to identify novel genes associated with both asthma pathogenesis (differentially expressed in the exposure-response study) and asthma susceptibility (genetically associated with asthma in a linkage/association study).

Patients with asthma and allergic rhinitis have long been known to have positive skin test responses to house dust. In the 1960's it was shown that the dust mite was the most important source of allergen in house dust. Techniques for growing dust mites in the laboratory enabled the preparation of dust mite allergen extracts. Identification of the major allergens of dust mite along with specific skin test methodology has resulted in standardized dust mite allergen extracts for diagnostic and therapeutic use. Numerous epidemiologic studies have demonstrated the importance of sensitization to dust mite as risk factors for asthma and allergic rhinitis symptoms.

Administration of dust mite by inhalation is considered investigational. However, numerous studies demonstrate the safety of allergen inhalation in well characterized subjects. A recent NHLBI/NIAID Workshop summarized evidence of the safety and utility of research bronchoprovocation and bronchoscopy studies in subjects with chronic airway diseases. Bronchoprovocation challenge has emerged as an important tool to understand the environmental factors involved in the asthmatic response. Airway hyperresponsiveness (AHR), an exaggerated bronchoconstrictor response to a variety of stimuli, is a prominent characteristic of asthma. Importantly, AHR to methacholine is correlated with symptoms and severity of disease. Although the mechanisms underlying AHR are poorly understood, it is believed to result, at least in part, from airway inflammation. Bronchoprovocation is a well-established method to detect and quantify AHR and to obtain insights into the mechanisms associated with this pathophysiologic entity. Increased airway response after allergen inhalation parallels the subsequent inflammatory reaction, suggesting that the allergen-induced inflammation has direct effects on mechanisms of airway responsiveness. Moreover, the techniques and applications of bronchoprovocation, both for testing nonspecific airway responsiveness and specific allergen challenge, have been well defined. Therefore it is evident that bronchoprovocation testing is considered useful and safe, and also likely to yield important insights into the pathogenesis of asthma.

Bronchoscopic airway sampling for investigational purposes has also yielded important insights regarding the pathogenesis of asthma and related airway disorders. Bronchoalveolar lavage (BAL) and endobronchial brush biopsies have emerged as the most widely used invasive research tools to assess inflammation and tissue remodeling in airway and interstitial lung diseases. Such procedures allow airway inflammatory and epithelial cells, proteins and other molecules of interest to be isolated in vivo in a manner that is critical to understanding the complex nature of asthma and other airway disorders. Numerous reports have attested to the safety of bronchoscopy including BAL and brush biopsy; these reports have been reviewed recently in a joint publication between the NHLBI and NIAID. So not only is bronchoscopic airway sampling important scientifically, but it is considered appropriate for research use in normal and asthmatic subjects.

The combination of bronchoprovocation and bronchoscopic airway sampling thus seems ideally suited to understand the complex host-environment interactions of asthma: the environmental stimulus response in a specified host could trigger a number of reactions that could be measured in the distal airways and airway epithelia.

ELIGIBILITY:
Inclusion Criteria:

* Allergic asthmatic, or nonallergic nonasthmatic
* Willing/able to give informed consent & adhere to visit/protocol schedules.
* Screening visit laboratory, C-Xray, EKG, results within normal limits
* Women of childbearing potential must have a negative serum pregnancy test
* Screening Pulmonary function testing above study criteria parameters

Exclusion Criteria:

* Systemic corticosteroid administration for asthma within the previous 90days
* Antibiotic administration within the previous 30 days.
* Viral respiratory infection within the previous 14 days.
* Allergen immunotherapy to House dust mite within the last 10 years
* History of severe asthma requiring intubation.
* Occupational exposure to hay or grain dust.
* Significant exposure history to cigarette smoke
* Past or present history of allergen immunotherapy to within the last 10 yrs
* Underlying illnesses that may result in altered lung function
* Students or employees under direct supervision by protocol investigators are ineligible
* Subjects allergic to medications used (or potentially used) in the study will be excluded.
* Subjects using aspirin will be excluded
* Subjects who abuse alcohol or illicit substances will be excluded
* Medication use other than for asthma, allergies or contraception
* Other medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements
* Nursing mothers
* Other investigational medication within the last 30 days

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-10; Primary Completion 2008-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Identify genes in airway epithelial and BAL cells that are differentially expressed following inhalation of house dust mite allergen among study subjects with allergic asthma and normal phenotypes. | 24 hours post challenge

CONTACTS AND LOCATIONS:
Overall Officials: John S Sundy, M.D., PhD., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States